CLINICAL TRIAL: NCT04731701
Title: Psychometric Validation of the Hemophilia Functional Ability Scoring Tool (Hemo-FAST)
Acronym: Hemo-FAST
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Kantar Health (Industry); Cerner Enviza (former Kantar Health) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Sobi.HAEM89-005
Record Dates: First submitted 2020-11-24; First posted 2021-02-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hemophilia Joint Health Score (HJHS) — Joint examination with Hemophilia Joint Health Score (HJHS)

SUMMARY:
The purpose of this study is to validate the newly developed Hemophilia Functional Ability Scoring Tool (Hemo-FAST), which is a fast and simple scoring in haemophilia able to assess patient-reported functional mobility.

DETAILED DESCRIPTION:
The purpose of this study is to validate the newly developed Hemophilia Functional Ability Scoring Tool (Hemo-FAST), which is a fast and simple scoring in haemophilia able to assess patient-reported functional mobility for adult haemophilia patients.

ELIGIBILITY:
Inclusion Criteria:A patient must fulfil the following criteria in order to be included in the study:

1. Age ≥18 years.
2. Diagnosis of haemophilia A or B.
3. Capable of completing the study Patient-Reported Outcome (PRO) questionnaires in French.
4. Signed informed consent.

Exclusion Criteria:

The presence of any of the following criteria will exclude a patient from inclusion in the study:

1. Joint replacement within last 6 months.
2. Patients with a non-resolved joint or muscle bleeding event at the enrolment visit or ≤ 7 days prior to the enrolment visit.
3. Patients with comorbid illnesses such as juvenile arthritis, muscular dystrophy, neurologic illness/cognitive impairment, or other illnesses that may independently affect HJHS and Hemo-FAST scores and/or limit the ability of the patient to participate in the study as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from 10-15 haemophilia treatment centres (HTCs) across France. The lower age limit of 18 years has been chosen because Hemo-FAST was developed to be used among the adult population. Age is an important contributor to the development of joint damage. Enrolment will therefore be targeted so that there will be similar numbers of patients enrolled across three age groups: 18-29, 30-44 and ≥ 45-years old.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Psychometric validation of the Hemophilia Functional Ability Scoring Tool (Hemo-FAST). | Baseline
  Statistical analysis to confirm the psychometric validation of the Hemo-FAST questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Swedish Orphan Biovitrum
Locations (16):
- France (16):
  - Swedish Orphan Biovitrum Clinical site, Paris, Cochin
  - Swedish Orphan Biovitrum Clinical site, Paris, Kremlin-Bicêtre
  - Swedish Orphan Biovitrum Clinical site, Besançon
  - Swedish Orphan Biovitrum Clinical site, Bordeaux
  - Swedish Orphan Biovitrum Clinical site, Brest
  - Swedish Orphan Biovitrum Clinical site, Caen
  - Swedish Orphan Biovitrum Clinical site, Clermont-Ferrand
  - Swedish Orphan Biovitrum Clinical site, Dijon
  - Swedish Orphan Biovitrum Clinical site, Lyon
  - Swedish Orphan Biovitrum Clinical site, Marseille
  - Swedish Orphan Biovitrum Clinical site, Nancy
  - Swedish Orphan Biovitrum Clinical site, Nantes
  - Swedish Orphan Biovitrum Clinical site, Rouen
  - Swedish Orphan Biovitrum Clinical site, Saint-Etienne
  - Swedish Orphan Biovitrum Clinical site, Strasbourg
  - Swedish Orphan Biovitrum Clinical site, Toulouse

IPD SHARING:
Plan to Share IPD: No